CLINICAL TRIAL: NCT01867983
Title: Comparative Effectiveness of Adding Weight Control to Smoking Cessation Quitlines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: SRI International (Industry); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DA031147 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Cigarette Smoking; Overweight; Obesity
Keywords: Tobacco cessation; Weight gain prevention
MeSH Terms: conditions — Cigarette Smoking; Overweight; Obesity; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Behavioral: Smoking cessation
  Interventions: Behavioral: Smoking cessation
- Simultaneous (Experimental): Behavioral: Weight gain prevention and smoking cessation
  Interventions: Behavioral: Weight gain prevention and smoking cessation
- Sequential (Experimental): Behavioral: Weight gain prevention and smoking cessation
  Interventions: Behavioral: Weight gain prevention and smoking cessation

INTERVENTIONS:
Behavioral: Weight gain prevention and smoking cessation — The two intervention groups will receive weight gain prevention either:
  Simultaneous: weight control treatment simultaneous with cessation treatment (5 proactive calls with a quit coach combined with weight coach/nutritionist followed by 5 'contact control calls'), or Sequential: weight control treatment added after cessation treatment (5 proactive calls with a quit coach followed by 5 weight coach/nutritionist calls). All three study arms will include a total of 10 phone counseling calls, interactive web, mailed support materials, access to nicotine replacement therapy (NRT) and unlimited participant initiated calls.
  Other Names: Tobacco cessation quitline; Weight management treatment
  Arms: Sequential; Simultaneous
Behavioral: Smoking cessation — The control group will receive cessation treatment calls (5 proactive calls with a quit coach followed by 5 contact control calls.
  Other Names: Tobacco cessation quitline
  Arms: Control

SUMMARY:
This randomized controlled trial compares the effectiveness for both smoking cessation and weight control of two alternative combined interventions offered via telephone quitline, as compared to standard of care quitline treatment addressing cessation alone. The interventions to be compared are cessation treatment alone versus cessation treatment combined with weight control treatment added either simultaneously or sequentially.

DETAILED DESCRIPTION:
Cigarette smoking and obesity are the leading causes of preventable morbidity and mortality in the U.S. Quitting smoking can lead to weight gain and obesity-related co-morbidities. Quitlines provide a natural population-based laboratory to test innovative approaches to help people quit smoking and control their weight. However, there is a lack of understanding of the effectiveness of intervening on both smoking and weight at the same time. Thus, we propose to test the impact on abstinence and weight control of adding an evidence-based weight control intervention simultaneously with or sequentially (following) cessation treatment via telephone quitlines.

This study, modeled on Co-I Dr. Bonnie Springs successful efficacy trial, is the first attempt to replicate the findings using widely available phone and web-based programs. The cessation program will be the effective and cost effective Quit For Life® quitline operated by Alere Wellbeing. The weight management program will be the Weight Talk program operated by Alere Wellbeing, also shown to be feasible, acceptable and effective in producing positive changes in weight, eating behaviors and physical activity. We will be using 5 calls from the Weight Talk program for the intervention content for the simultaneous and sequential arms.

The proposed randomized controlled trial compares the effectiveness for both smoking cessation and weight control of two alternative combined interventions offered via telephone quitline, as compared to standard of care quitline treatment addressing cessation alone. The interventions to be compared are cessation treatment alone versus cessation treatment combined with weight control treatment added either simultaneously or sequentially. We propose to recruit 2550 smokers who call a quitline and randomly assign them to one of three groups: (a) Standard Care (STD): cessation treatment calls (5 proactive calls with a quit coach followed by 5 contact control calls); (b) Simultaneous: weight control treatment simultaneous with cessation treatment (5 proactive calls with a quit coach combined with weight coach/nutritionist followed by 5 'contact control calls'), or (c) Sequential: weight control treatment added after cessation treatment (5 proactive calls with a quit coach followed by 5 weight coach/nutritionist calls). All three interventions include a total of 10 phone counseling calls, interactive web, mailed support materials, access to nicotine replacement therapy (NRT) and unlimited participant-initiated calls.

Significance: This study is novel. Combining two phone/web based behavior change programs together has never been tested. A cost-effective, population-based strategy for delivering a combined smoking cessation and weight control intervention stands to make a significant impact. The option of new telephone counseling that helps smokers quit and control their weight could encourage smokers to call quitlines who otherwise might not because they are concerned about gaining weight. Combined smoking and weight treatment could also increase abstinence rates over current best-practice treatment and do so without weight gained its adverse consequences. Moreover, if effective, the intervention could rapidly be disseminated to the 500,000 smokers who use quitlines annually in the U.S., a large proportion of whom are obese.

ELIGIBILITY:
Inclusion Criteria:

* Participating Client
* Not Re-Enrolling
* USA Resident
* Wants to quit in the next 30 days
* Use Cigarettes (other types ok, but must use cigarettes)
* 18 years or older
* Speak English
* Provide Phone
* Provide Email Address
* Use 10 cigarettes per day or more
* BMI of 18.5 or above
* No history of anorexia or bulimia

Exclusion Criteria:

* Pregnant or Planning Pregnancy within 3 months
* Diabetic
* Previous weight loss surgery or planning weight loss surgery in next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2540 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence tobacco abstinence | 6 months
Change in weight | 6 months

SECONDARY OUTCOMES:
Other abstinence effectiveness (7-day, continuous abstinence, reduction in amount) | 6 and 12 months
Cost-effectiveness (cost per quit) | 6 and 12 months
Weight control cost-effectiveness (cost per pound not gained) | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Terry Bush, PHD, Principal Investigator — Consumer Wellness Solutions
Locations (1):
- Alere Wellbeing, Seattle, Washington, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Javitz HS, Bush TM, Lovejoy JC, Torres AJ, Wetzel T, Wassum KP, Tan MM, Alshurafa N, Spring B. Six Month Abstinence Heterogeneity in the Best Quit Study. Ann Behav Med. 2019 Nov 9;53(12):1032-1044. doi: 10.1093/abm/kaz014. PMID 31009528
- [Derived] Bush T, Lovejoy J, Javitz H, Torres AJ, Wassum K, Tan MM, Spring B. Simultaneous vs. sequential treatment for smoking and weight management in tobacco quitlines: 6 and 12 month outcomes from a randomized trial. BMC Public Health. 2018 May 31;18(1):678. doi: 10.1186/s12889-018-5574-7. PMID 29855294
- [Derived] Bush T, Lovejoy J, Javitz H, Magnusson B, Torres AJ, Mahuna S, Benedict C, Wassum K, Spring B. Comparative effectiveness of adding weight control simultaneously or sequentially to smoking cessation quitlines: study protocol of a randomized controlled trial. BMC Public Health. 2016 Jul 22;16:615. doi: 10.1186/s12889-016-3231-6. PMID 27443485